CLINICAL TRIAL: NCT01012102
Title: An Open Label, Parallel Group, Randomized Phase I Study of Biological Activity, Safety, Tolerability, and Clinical Activity of Different Dose Levels of EMD 640 744 in Montanide ISA 51 VG Administered in Subjects With Advanced Solid Tumors
Brief Title: EMD 640 744 in Montanide ISA 51 VG Administered in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200032-001
Record Dates: First submitted 2009-10-20; First posted 2009-11-11 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2011-10

CONDITIONS: Advanced Solid Tumors
Keywords: EMD 640744; Montanide; Advanced solid tumours
MeSH Terms: interventions — montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): EMD 640744 30μg and Montanide® ISA 51 VG
  Interventions: Biological: EMD 640744; Other: Montanide ISA 51 VG
- Group 2 (Experimental): EMD 640744 100μg and Montanide® ISA 51 VG
  Interventions: Biological: EMD 640744; Other: Montanide ISA 51 VG
- Group 3 (Experimental): EMD 640744 300μg and Montanide® ISA 51 VG
  Interventions: Biological: EMD 640744; Other: Montanide ISA 51 VG

INTERVENTIONS:
Biological: EMD 640744 — EMD 640744 30μg, weekly in initiation phase and monthly in maintenance phase (in combination with Montanide® ISA 51 VG)
  Arms: Group 1
Biological: EMD 640744 — EMD 640744 100μg, weekly in initiation phase and monthly in maintenance phase (in combination with Montanide® ISA 51 VG)
  Arms: Group 2
Biological: EMD 640744 — EMD 640744 300μg, weekly in initiation phase and monthly in maintenance phase (in combination with Montanide® ISA 51 VG)
  Arms: Group 3
Other: Montanide ISA 51 VG — Adjuvant. Montanide® ISA 51 VG, weekly in initiation phase and monthly in maintenance phase (in combination with EMD 640744 30ug)
  Arms: Group 1
Other: Montanide ISA 51 VG — Adjuvant. Montanide® ISA 51 VG, weekly in initiation phase and monthly in maintenance phase (in combination with EMD 640744 100ug)
  Arms: Group 2
Other: Montanide ISA 51 VG — Adjuvant. Montanide® ISA 51 VG, weekly in initiation phase and monthly in maintenance phase (in combination with EMD 640744 300ug)
  Arms: Group 3

SUMMARY:
To compare 3 doses of EMD 640744 administered by subcutaneous injection in combination with Montanide® ISA 51 VG with regard to immunological efficacy.

The primary target variable is the immune response as assessed by ELISPOT before and until week 17 after vaccination with EMD 640744 in Montanide® ISA 51 VG.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Signed written informed consent
* Histologically or cytologically documented metastatic or locally advanced survivin-expressing solid tumor for which no established therapy exists
* Disease must be measurable by RECIST criteria or evaluable by clinical, radiographic, or laboratory criteria established for the given tumor entity
* Expressing at least one of the following HLA alleles:HLA-A1,-A2,-A3,-A24, and -B7 assessed by HLAgenotyping
* ECOG performance status of ≤1, estimated life expectancy of at least 3 months
* Adequate hematological function defined by WBC ≥3 x 10x9/L, lymphocyte count ≥0.5 x 10x9/L, hemoglobin ≥10 g/dL, platelet count ≥100 x 10x9/L
* Adequate blood coagulation parameters defined as aPTT and INR ≤ 1.5 x ULN
* Adequate renal function defined by a serum creatinine ≤2 x ULN
* Adequate hepatic function defined by total bilirubin ≤2 x ULN and AST and ALT levels ≤2.5 x ULN (in subjects with liver metastases ≤5 x ULN)
* Effective contraception for female and male subjects if the risk of conception exists

Exclusion Criteria:

* Treatment in another clinical study within the past 30 days prior to the first administration of study treatment
* Previous treatment with an investigational anticancer vaccine
* Requirement of concurrent treatment with a nonpermitted drug
* Active significant autoimmune disease (with the exception of vitiligo)
* Receipt of allogeneic stem cell transplantation
* Significant acute or chronic infections (e.g. viral hepatitis, HIV)
* Primary brain tumors and brain metastases (with the exception of brain metastases that are stable after irradiation or surgically resected brain metastases if subjects have been asymptomatic for ≥6 months)
* Rapidly progressive disease (e.g. tumor lysis syndrome)
* Radiotherapy, chemotherapy, surgery (excluding prior diagnostic biopsy), immunotherapy or any investigational drug within 30 days before the start of study treatment
* Pregnancy or lactation
* Active drug or alcohol abuse
* Known hypersensitivity to the study treatment or any of its components
* Any significant disease that, in the Investigator's opinion, should exclude the subject from the study; for questions about this criterion, the Investigator should contact the sponsor.
* Persisting toxicity related to prior therapy ≥grade 2 National Cancer Institute-Common Terminology Criteria For Adverse Events version 3.0
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To compare 3 doses of EMD 640744 administered by subcutaneous injection in combination with Montanide® ISA 51 VG with regard to immunological efficacy | 1-4 weeks

SECONDARY OUTCOMES:
To assess the safety and tolerability of different doses of EMD 640744 in Montanide® ISA 51 VG in terms of laboratory parameters and adverse event profile. | 3 months
To assess the clinical efficacy in terms of the overall response, progression-free survival time, and survival time. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Peter Marschner, MD, Study Director — Merck KGaA, Darmstadt

REFERENCES:
- [Result] Lennerz V, Gross S, Gallerani E, Sessa C, Mach N, Boehm S, Hess D, von Boehmer L, Knuth A, Ochsenbein AF, Gnad-Vogt U, Zieschang J, Forssmann U, Woelfel T, Kaempgen E. Immunologic response to the survivin-derived multi-epitope vaccine EMD640744 in patients with advanced solid tumors. Cancer Immunol Immunother. 2014 Apr;63(4):381-94. doi: 10.1007/s00262-013-1516-5. Epub 2014 Feb 2. PMID 24487961